CLINICAL TRIAL: NCT06396377
Title: Interest of the Reborn® Doll as a Therapeutic Object in the Care of Residents With Alzheimer's Disease or a Related Disorder : Pilote Study
Brief Title: Interest of the Reborn® Doll as a TO in the Care of Residents With Alzheimer's Disease or a Related Disorder
Acronym: PROTMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RBHP 2023 MARTIN; 2023-A00383-42 (Other: ANSM)
Record Dates: First submitted 2024-04-05; First posted 2024-05-02 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Dementia Alzheimers
Keywords: Alzheimer; Reborn doll; agitation; behavioural disorders; cognitive disorders
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Mental Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: randomized parallel-arm trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): If the resident is randomized to the control group, the resident will not receive a reborn®doll. The investigating team will observe the resident's behavior as if he or she were receiving a doll.
- Reborn doll (Experimental): The investigating team will give the Reborn®doll to the resident, during a 45-minute to 1-hour workshop, twice a week for 3 weeks. The OTs, wrapped in a blanket, are presented to the residents by a member of the investigative team trained in reborning , in the resident's room. If the resident is not in his/her room, he/she will be taken back to receive his/her doll. In the case of double rooms, it will be necessary to assess whether or not to leave the room-mate in the room, in order to limit the loss of reference points for the resident concerned by the study. The caregiver lets the resident appropriate and recognize the OT, so that he or she can find meaning in it and awaken his or her sensory memory.In total, the patient will be exposed to OT 6 times.
  Interventions: Device: Reborn doll (Therapeutic object - OT)

INTERVENTIONS:
Device: Reborn doll (Therapeutic object - OT) — If the resident is randomized to the intervention group, the investigating team will give the Reborn®doll to the resident, during a 45-minute to 1-hour workshop, twice a week for 3 weeks. The OTs, wrapped in a blanket, are presented to the residents by a member of the investigative team trained in reborning , in the resident's room. If the resident is not in his/her room, he/she will be taken back to receive his/her doll. In the case of double rooms, it will be necessary to assess whether or not to leave the room-mate in the room, in order to limit the loss of reference points for the resident concerned by the study. The caregiver lets the resident appropriate and recognize the OT, so that he or she can find meaning in it and awaken his or her sensory memory.In total, the patient will be exposed to OT 6 times.
  Arms: Reborn doll

SUMMARY:
The primary objective of this study is to evaluate the benefits of the Reborn®doll as an OT for the care of residents with Alzheimer's disease or related disorders, by assessing the frequency of resident agitation.

The secondary objectives are to study the frequency of treatments, evaluate the average time of exposure to the Reborn® doll, study the behavior of the residents, study the interest of this therapeutic workshop, thanks to an evaluation grid and finally study the repercussions of this OT on the nursing staff.

DETAILED DESCRIPTION:
Dementia affects 50 million people worldwide, and this number is set to continue rising as the population ages. Indeed, the World Health Organization (WHO) expects this number to reach 82 million by 2030. At present, there is no cure for dementia. In order to limit the need for drug treatments for dementia-related symptoms (agitation, aggression), non-drug treatments can be used to improve residents' lives and soothe them. In the late 1960s, researchers turned their attention to non-medication therapies (snozelen concept, animal mediation, calinotherapy, Tovertafel, Carpe Diem, doll'therapy).

This doll is used by caregivers to calm anxiety attacks, aggression or apathy in residents with MND. The doll helps to calm the elderly by focusing them on an object. Several studies have shown that residents are calmed and feel valued by taking care of the doll. This also helps to avoid physical or chemical restraints, as well as the use of drug therapies in cases of agitation. Reborn® dolls are an evolution of Doll'therappy.

ELIGIBILITY:
Inclusion Criteria:

* Resident aged 65 and over
* Moderate to severe cognitive impairment diagnosed using the NPI-ES scale
* Behavioral disorders (agitation, aggression, anxiety, apathy) assessed using the NPI-ES scale
* Covered by a social security plan
* Written consent of representative (tutor/ curator/trusted person)

Exclusion Criteria:

* Resident or representative refusing to participate
* Resident under judicial protection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Episodes of resident agitation using the Cohen Mansfield scale | During the study period (4 weeks)
  The number of episodes of agitation will be collected weekly by the nursing assistant or nurse in charge of monitoring, by compiling the events reported on a resident monitoring document with the time of recording.
  The characterization of these episodes should correspond to one of the items on the Cohen Mansfield scale. Two consecutive episodes cannot be counted if they are less than one hour apart (and will therefore be counted as a single event). Follow-up should be strictly identical, whether the resident belongs to the intervention group or the control group.

SECONDARY OUTCOMES:
Factors that can affect doll benefits: gender, age, pathology, Charlson Comorbidity Index, doll identifier. | Inclusion
Drug treatments | During the study period (4 weeks)
  Medication during study period (name/posology) if applicable (daily record)
Average exposure time to Reborn®dolls | During the study period (4 weeks)
  Average exposure time to Reborn®dolls in minutes
Therapeutic evaluation scale | During the study period (4 weeks)
  Therapeutic evaluation grid only on days when residents are in possession of the OT on the Crossway computerized file
Quality of working life questionnaire | During the study period (4 weeks)
  Quality of working life questionnaire to be completed by nursing staff on the Friday of the observation week, and on the last Friday (last day of the study).
Resident behavior following OT withdrawal | During the study period (4 weeks)
  Resident behavior following OT withdrawal (for experimental group). Observation of the care team.
Resident behavior after OT exposure | During the study period (4 weeks)
  Resident behavior after OT exposure. Observation of the care team.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Afonso, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France